CLINICAL TRIAL: NCT00642798
Title: An Open-Label, Single- & Multiple-Dose Study to Investigate the Pharmacokinetics of Sitagliptin 100 mg in Healthy Chinese Adult Subjects
Brief Title: An Open-Label, Single- & Multiple-Dose Study to Investigate the Pharmacokinetics of Sitagliptin 100 mg in Healthy Chinese Adult Subjects (0431-108)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0431-108; 2008_002
Record Dates: First submitted 2008-03-07; First posted 2008-03-25 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes Mellitus Non-insulin-dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

INTERVENTIONS:
Drug: sitagliptin phosphate — Sitagliptin 100mg once daily on Day 1 for single dose, and once daily on Day4-9 for multiple dose.
  Other Names: Januvia™; MK0431

SUMMARY:
To support the registration of sitagliptin 100mg in china.

ELIGIBILITY:
Inclusion Criteria:

* Subject Has Been A Nonsmoker And/Or Has Not Used Nicotine Or Nicotine-Containing Products For At Least Approximately 6 Months; Subjects Who Have Discontinued Smoking Or The Use Of Nicotine/Nicotine Containing Products For At Least Approximately 3 Months May Be Enrolled In The Study At The Discretion Of The Investigator
* Subject Has No Clinically Significant Abnormality On Electrocardiogram (Ecg) Performed At The Prestudy (Screening) Visit And/Or Prior To Administration Of The Initial Dose Of Study Drug
* Subject Is Judged To Be In Good Health Based On Medical History, Physical Examination, Vital Sign Measurements, And Laboratory Safety Tests Performed At The Prestudy (Screening) Visit And/Or Prior To Administration Of The Initial Dose Of Study Drug
* Subject Is Male Or Female 18 To 45 Years Of Age At The Prestudy (Screening) Visit. Female Subjects Of Reproductive Potential Must Demonstrate A Serum Beta-Hcg Level Consistent With The Nongravid State At The Prestudy (Screening) Visit And Agree To Use (And/Or Have Their Partner Use) Two Acceptable Methods Of Birth Control Beginning At Least 2 Weeks Prior To Administration Of The First Dose Of Study Drug, Throughout The Study (Including Washout Intervals Between Treatment Periods/Panels) And Until At Least 2 Weeks After Administration Of The Last Dose Of Study Drug In The Last Treatment Period. Acceptable Methods Of Birth Control Are: Abstinence, Intrauterine Device (Iud), Diaphragm, Spermicides, Cervical Cap, Contraceptive Sponge, And Condoms
* Subject Is Of Chinese Descent With All 4 Biological Grandparents Born In China And Of Chinese Descent
* Subject Is Willing To Comply With The Study Restrictions
* Subject Understands The Study Procedures And Agrees To Participate In The Study By Giving Written Informed Consent
* The Subject Has A Body Mass Index (BMI) Between 19 And 24 Kg/M2 And The Body Weight Is More Than 50 Kg At The Prestudy (Screening) Visit.

Exclusion Criteria:

* Subject Consumes Excessive Amounts Of Alcohol, Defined As Greater Than 3 Glasses Of Alcoholic Beverages (1 Glass Is Approximately Equivalent To: Beer [284 Ml/10 Ounces],Wine [125 Ml/4 Ounces], Or Distilled Spirits [25 Ml/1 Ounce]) Per Day. Subjects That Consume 4 Glasses Of Alcoholic Beverages Per Day May Be Enrolled At The Discretion Of The Investigator
* Subject Consumes Excessive Amounts, Defined As Greater Than 6 Servings (1 Serving Is Approximately Equivalent To 120 Mg Of Caffeine) Of Coffee, Tea, Cola, Or Other Caffeinated Beverages Per Day
* Subject Has A History Of Any Illness That, In The Opinion Of The Study Investigator, Might Confound The Results Of The Study Or Poses An Additional Risk To The Subject By Their Participation In The Study
* Subject Has A History Of Neoplastic Disease.
* Subject Has A History Of Significant Multiple And/Or Severe Allergies, Or Has Had An Anaphylactic Reaction Or Significant Intolerability To Prescription Or Non-Prescription Drugs Or Food
* Subject Has A History Of Stroke, Chronic Seizures, Or Major Neurological Disorder
* Subject Has An Estimated Creatinine Clearance Of <=80 Ml/Min Based On The Cockcroft-Gault Equation
* Subject Has Had Major Surgery, Donated Or Lost 1 Unit Of Blood (Approximately 500 Ml) Or Participated In Another Investigational Study Within 4 Weeks Prior To The Prestudy (Screening) Visit
* Subject Is A Nursing Mother
* Subject Is Currently A Regular User (Including Recreational Use)Of Any Illicit Drugs Or Has A History Of Drug (Including Alcohol) Abuse Within Approximately 6 Months
* Subject Is Mentally Or Legally Incapacitated, Has Significant Emotional Problems At The Time Of Prestudy (Screening) Visit Or Expected During The Conduct Of The Study Or Has A History Of A Clinically Significant Psychiatric Disorder Over The Last 5 To 10 Years.Subjects Who Have Had Situational Depression May Be Enrolled In The Study At The Discretion Of The Investigator
* Subject Is Unable To Refrain From Or Anticipates The Use Of Any Medication, Including Prescription And Non-Prescription Drugs Or Herbal Remedies (Such As St. John Wort[Hypericum Perforatum]) Beginning Approximately 2 Weeks (Or 5 Half-Lives) Prior To Administration Of The Initial Dose Of Study Drug, Throughout The Study (Including Washout Intervals Between Treatment Periods), Until The Post-study Visit
* Subject Is Under The Age Of Legal Consent
* There Is Any Concern By The Investigator Regarding The Safe Participation Of The Subject In The Study Or For Any Other Reason, The Investigator Considers The Subject Inappropriate For Participation In The Study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of sitagliptin after administration of single and multiple 100-mg doses of sitagliptin to healthy chinese adult subjects. | Duration of Trial

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC